CLINICAL TRIAL: NCT03942926
Title: The Efficacy and Safety of Sirolimus for Plastic Bronchitis：a Pilot Study
Brief Title: The Efficacy and Safety of Sirolimus for Plastic Bronchitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: North-China Pharmaceutical Company, China (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PB1
Record Dates: First submitted 2019-05-05; First posted 2019-05-08 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Plastic Bronchitis
Keywords: plastic bronchitis; sirolimus
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Intervention Model Description: Ten lymphatic bronchitis patients are planned to be recruited for the study. Sirolimus will be administered for 6 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sirolimus (Experimental): Patients in sirolimus group will receive sirolimus for 6 months.
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Patients will receive sirolimus for 6 months.
  Other Names: rapamycin

SUMMARY:
There is no confirmed drug therapy for plastic bronchitis. The study wish to test the effectiveness and safety of sirolimus (rapamycin) in patients with lymphatic plastic bronchitis.

DETAILED DESCRIPTION:
Plastic bronchitis is a rare respiratory disorder characterized by formation of gelatinous or rigid cast of bronchial tree. Confirmed drug therapy for plastic bronchitis is lacking. Recently, part of plastic bronchitis has been found to have dysfunction of lymphatic circulation in the lung. Pulmonary lymphatic perfusion syndrome (PLPS) is regarded as a major mechanism of lymphatic plastic bronchitis. Sirolimus (rapamycin) has not been studied in plastic bronchitis, however, it has been shown effective in several lymphatic disorders, such as lymphangioleiomyomatosis, generalized lymphatic anomaly (GLA) including lymphangiomatosis, etc. We wish to test the effectiveness of sirolimus in lymphatic plastic bronchitis.

ELIGIBILITY:
Inclusion Criteria:

* plastic bronchitis
* pulmonary lymphatic perfusion syndrome demonstrated on 68Ga-NEB positron emission tomography (PET)

Exclusion Criteria:

* Pregnancy and breastfeeding
* Severe cardiovascular, hepatic and renal dysfunction
* allergy to sirolimus or 68Ga-NEB

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-05-06 (Estimated); Primary Completion 2020-05-05 (Estimated); Study Completion 2020-05-05 (Estimated)

PRIMARY OUTCOMES:
changes of pulmonary lymphatic perfusion distribution | 6 months
  quantitatively measured with 68Ga-NEB positron emission tomography (PET) at baseline and the end of study
changes of coughing score | 6 months
  measured by coughing VAS score (0-10) at baseline, 3 months and the end of study

SECONDARY OUTCOMES:
changes of pulmonary function (FEV1, FVC) | 6 months
  measured by spirometry at baseline, 3 months and the end of study
changes of six minutes walking distance | 6 months
  measured by six minutes walking test at baseline, 3 months and the end of study
change of health-related quality of life | 6 months
  measure by St George Respiratory Questionnaire at baseline, 3 months and the end of study
changes of breathlessness score | 6 months
  measured by Borg scale (0-10) at baseline, 3 months and the end of study
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 6 months
  Common Terminology Criteria for Adverse Events (CTCAE) was used to collect adverse effects at baseline and through study completion

CONTACTS AND LOCATIONS:
Overall Officials: Kai-Feng Xu, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The protocol and clinical study report will be shared.
Supporting Information: Study Protocol, CSR
Time Frame: Data will be shared between time of completion of the study and time of publication of the study.
Access Criteria: contact principle investigator Dr Kai-Feng Xu via xukf@pumch.cn